CLINICAL TRIAL: NCT05879445
Title: Causes, Complications and Outcomes of Severe Acute Liver Disease Cases Admitted to Intensive Care Units
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdallah Hussein Kamel Ibrahim, Resident Physician, Assiut University
Other Study IDs: Severe ALD in intensive care
Record Dates: First submitted 2023-04-07; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Acute Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute liver failure (ALF) is a potentially fatal complication of severe hepatic illness resulting from various causes. In a clinical setting, severe hepatic injury is usually recognized by the appearance of jaundice, encephalopathy and coagulopathy.

The term acute liver failure (ALF) is frequently applied as a generic expression to describe patients presenting with or developing an acute episode of liver dysfunction.

Cerebral edema is very common in patients with acute liver failure and encephalopathy.

Acute liver failure (ALF) has Less common aetiologies include viral hepatitis, drug-induced liver injury, pregnancy-induced liver failure and autoimmune hepatitis.

Survival for patients with ALF has steadily improved over the last few decades. Acute liver failure (ALF) is defined as sever acute liver injury with encephalopathy and impairment of synthetic function (INR ˃1.5) in a patient without pre-existing cirrhosis or liver disease.

Acute liver failure (ALF) and acute on chronic liver Failure (ACLF) are conditions frequently encountered in the ICU and are associated with high mortality.

DETAILED DESCRIPTION:
The main objectives of this observational study are:

1. To evaluate cases of (ALF) and (ACLF) according to guidelines.
2. To determine most likely causes of disease in a patient of each age.
3. To determine complications of disease.
4. Assesment of mortality and morbidity rates.
5. Assessment of in-hospital and six month follow up outcomes according to guidelines.

Participants (or their designated contact persons) will be contacted over the phone for either a telephone interview or a follow-up visit in the outpatient clinics, whichever feasible and possible.

All patients presented with severe acute liver disease, acute liver failure (ALF) and acute on chronic liver disease (ACLF).

1. Inclusion criteria:

   1. reduced conscious state
   2. Jaundice with abnormal liver function tests, especially elevations in amino acid transferase levels more than 25 times the upper limit of normal
   3. Coagulopathy
   4. Multiorgan failure
2. Exclusion criteria:

Patients with these criteria will be excluded:

1. Patients with known cardiac cirrhosis.
2. Patients with known pre-existing renal disease

   * Study tools

All patients will be subjected to:

1. Thorough history taking (History of previous renal disease, severe co-morbidity, malignancy, …).
2. Thorough clinical examination

   1. Vital signs.
   2. General examination.
   3. Systemic examination:

      * Chest examination.
      * Cardiac examination.
      * Abdominal examination.
      * Neurological examination.
3. Imaging

   1. Abdominal ultrasound with especial comment on kidneys and intra-abdominal fluid.
   2. Chest x-ray
   3. Echocardiography
4. Laboratory investigations

   1. Liver function tests: alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), serum bilirubin, prothrombin time (PT) and albumin.

      Before and after end of treatment.
   2. Serum creatinine:

      Before and after end of treatment
   3. Urine analysis:

      Before and after end of treatment
   4. Albumin creatinine ratio:

   Before and after end of treatment
5. Measuring body weight Before and after end of treatment
6. Special scores (CLIF-SOFA /CLIF-C OFs /DF /ABIC /GAHS /MELD /MELD-Na /CHILD)

ELIGIBILITY:
Inclusion Criteria:

1. reduced conscious state
2. Jaundice with abnormal liver function tests, especially elevations in amino acid transferase levels more than 25 times the upper limit of normal
3. Coagulopathy
4. Multiorgan failure

Exclusion Criteria:

1. Patients with known cardiac cirrhosis.
2. Patients with known pre-existing renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presented with severe acute liver disease, acute liver failure (ALF) and acute on chronic liver disease (ACLF).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Liver function in individuals with ALF admitted to intensive care unit. | 2 weeks after admission to intensive care unit
  Measuring serum alanine transaminase (ALT) level, serum aspartate transaminase (AST) level, serum alkaline phosphatase (ALP) level, serum gamma-glutamyl transferase (GGT) level.
Assessment of kidney function in individuals with ALF admitted to intensive care unit. | 2 weeks after admission to intensive care unit
  Measuring serum creatinine level
Assessment of fluid overload in individuals with ALF admitted to intensive care unit. | 2 weeks after admission to intensive care unit
  Measuring body weight.

SECONDARY OUTCOMES:
Mortality rates | 2 weeks after admission to intensive care unit
  Assessment of mortality rates in individuals with ALF admitted to intensive care unit.
Morbidity rates | 2 weeks after admission to intensive care unit
  Assessment of morbidity rates in individuals with ALF admitted to intensive care unit..